CLINICAL TRIAL: NCT07107464
Title: Subcrestal Placement of PRAMA Implants With Convergent Neck Incorporating Ultrathin Threaded Microsurface: A Randomized Controlled Clinical Trial
Brief Title: Subcrestal vs Juxtacrestal PRAMA Implants With Variable Necks
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ARDEC Academy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/02
Record Dates: First submitted 2025-07-19; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Edentulism; Dental Implantation, Endosseous; Marginal Bone Loss; Periimplant Bone Loss
Keywords: edentulism; dental implants; Peri-Implant Bone Loss; Subcrestal Implant Placement; One-Piece Implants; Implant Neck Design; Convergent Implant Neck

STUDY DESIGN:
Intervention Model Description: Split-mouth randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Allocation concealment is ensured via sealed opaque envelopes opened at the time of surgery. The surgeon is blinded to group assignment until after flap elevation, and the prosthetic team is unaware of crown design assignment until delivery. The outcomes assessor responsible for radiographic, CBCT, and 3D volumetric evaluations remains blinded to treatment allocation throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short Neck Implant - Crestal Placement (Experimental): Participants in this arm receive one-piece dental implants with a short transmucosal neck (1.8 mm total height, hyperbolic convergent shape) placed at the level of the bone crest (crestal placement). The implant features a ZirTi surface and Ultrathin Threaded Microsurface across the entire neck.
  Interventions: Device: Short Neck Implant - Crestal Placement
- Standard Neck Implant (1 mm Subcrestal Placement) (Experimental): Participants in this arm receive one-piece dental implants with a standard transmucosal neck (0.8 mm cylindrical plus 2.0 mm convergent portion) placed 1 mm below the bone crest. The implant surface includes micro-threads throughout the neck to promote tissue stability.
  Interventions: Device: Standard Neck Implant - 1 mm Subcrestal Placement
- Long Neck Implant (2 mm Subcrestal Placement) (Experimental): Participants in this arm receive one-piece dental implants with a long transmucosal neck (0.8 mm cylindrical plus 3.0 mm convergent portion) placed 2 mm below the bone crest. This arm tests the effect of deeper placement combined with extended neck geometry.
  Interventions: Device: Long Neck Implant - 2 mm Subcrestal Placement

INTERVENTIONS:
Device: Short Neck Implant - Crestal Placement — A one-piece endosseous dental implant with a 1.8 mm short convergent neck, placed at the bone crest. Implant used: PRAMA implant (Sweden & Martina, Italy) with UTM surface treatment.
  Arms: Short Neck Implant - Crestal Placement
Device: Standard Neck Implant - 1 mm Subcrestal Placement — A one-piece endosseous dental implant with a standard-length neck (2.8 mm total; 0.8 mm cylindrical + 2 mm convergent), placed 1 mm subcrestally. Implant used: PRAMA implant (Sweden & Martina, Italy) with UTM surface.
  Arms: Standard Neck Implant (1 mm Subcrestal Placement)
Device: Long Neck Implant - 2 mm Subcrestal Placement — A one-piece endosseous dental implant with a long transmucosal neck (3.8 mm total; 0.8 mm cylindrical + 3 mm convergent), placed 2 mm subcrestally. Implant used: PRAMA implant (Sweden & Martina, Italy) with UTM surface.
  Arms: Long Neck Implant (2 mm Subcrestal Placement)

SUMMARY:
The goal of this clinical trial is to understand how different implant neck designs and placement depths affect the surrounding bone and peri-implant tissue (the tissue around a dental implant) in adults who need implants in the back areas of the mouth (molars and premolars). The main questions it aims to answer are:

Does placing implants deeper under the bone crest (subcrestally) help preserve more bone and peri-implant tissue over time? Do implants with longer, conical necks and micro-threaded surfaces result in more stable peri-implant tissue than implants with shorter necks? Researchers will compare three types of one-piece dental implants with different neck heights (short, standard, and long), placed at different depths in the jawbone, to determine which combination better maintains bone and peri-implant tissue levels.

Participants will:

Receive two dental implants in the posterior upper or lower jaw Be randomly assigned to one of three groups depending on implant neck design and placement depth Undergo implant surgery using a digital workflow, with healing over three months Be rehabilitated with custom zirconia bridges Return for regular clinical and imaging checkups over a period of at least 3 years This study aims to generate evidence that helps clinicians choose implant designs and techniques that promote long-term peri-implant tissue health.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the impact of different transmucosal neck configurations and vertical placement levels of one-piece dental implants on peri-implant hard and soft tissue stability over time. The trial specifically focuses on the PRAMA implant system (Sweden & Martina, Italy), which incorporates a ZirTi surface and a convergent neck design with an Ultrathin Threaded Microsurface (UTM). These implants are designed to optimize tissue integration and minimize marginal bone loss.

The study explores how subcrestal versus crestal placement of the rough-to-smooth transition, combined with variable neck lengths, influences peri-implant tissue outcomes under functional loading in posterior edentulous sites. Three types of PRAMA implants will be compared:

Short neck (1.8 mm total length with hyperbolic convergent shape)

Standard neck (0.8 mm cylindrical plus 2.0 mm convergent portion)

Long neck (0.8 mm cylindrical plus 3.0 mm convergent portion)

Each patient will receive two implants to support a 2- or 3-unit prosthetic bridge. The neck design determines the depth of implant placement:

Short group: coronal rough surface margin placed at bone crest (crestal placement)

Standard group: 1 mm subcrestal placement

Long group: 2 mm subcrestal placement

The trial adopts a parallel design, with a sample size of 30 patients (10 per group), allowing for adequate power while considering possible dropouts. Randomization will be performed electronically and concealed in opaque envelopes until surgery. Blinding is partially feasible, especially for radiographic and digital analysis where treatment allocation is masked.

Surgical procedures will be standardized using a fully digital workflow. Implants will be placed in healed sites without the need for bone grafting. Healing will be non-submerged using appropriate healing abutments. After three months, definitive zirconia bridges will be installed, and patients will be enrolled in a maintenance protocol.

In addition to comparing the impact of different neck designs and placement depths, the prosthetic crowns will be designed with two distinct emergence profiles: one simulating a natural root form extending apically, and the other adapted to the mucosal margin. This design will allow for the assessment of volumetric tissue adaptation based on prosthetic contour.

Primary outcomes will include longitudinal changes in marginal bone height evaluated through standardized periapical radiographs, CBCT, and digital scans. Secondary outcomes include:

Volumetric soft tissue changes assessed using superimposed 3D models derived from intraoral scans.

Comparison of tissue responses between the two crown designs (root-form vs. standard emergence).

Clinical parameters such as probing depth, plaque index, and bleeding on probing at designated follow-ups.

Radiographic and volumetric measurements will be performed by calibrated, blinded examiners. Imaging will be taken at baseline (prosthesis delivery), 6 months, and annually up to 3 years. Analytical methods include ANOVA or Kruskal-Wallis tests based on data distribution, with appropriate post-hoc comparisons and a significance level set at p < 0.05.

This study is expected to contribute relevant clinical data to the ongoing discussion around subcrestal implant placement and the role of implant macro- and micro-geometry in maintaining peri-implant tissue health.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21 years or older.
* Presence of an edentulous area in the posterior maxilla or mandible (premolar or molar region) that allows the placement of two dental implants.
* Alveolar bone height sufficient to permit implant insertion with a minimum depth of 6 mm, and total implant length of at least 10 mm.
* Indication for implant-supported prosthetic restoration (2- or 3-unit fixed dental bridge).
* Good general health with no contraindications for oral surgical procedures.
* Not pregnant at the time of screening.
* Willingness and ability to sign written informed consent and comply with study procedures.

Exclusion Criteria:

* Presence of uncontrolled systemic disease (e.g., diabetes, cardiovascular disorders, immunosuppression).
* History of chemotherapy or radiotherapy to the head or neck region.
* Heavy smokers (defined as >10 cigarettes per day)
* Previous bone regeneration or grafting procedures at the target implant site.
* Use of medications known to interfere with bone metabolism (e.g., bisphosphonates, corticosteroids).
* Poor oral hygiene or active periodontal disease that may compromise implant success.

-Known allergy or hypersensitivity to implant materials used in the study-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Peri-Implant Bone Height Over Time | Baseline (prosthesis delivery), 6 months, and annually up to 3 years post-loading
  Vertical changes in marginal bone level from the implant-abutment junction to the first bone-to-implant contact (BIC) at mesial and distal aspects, measured on standardized periapical radiographs, CBCT, and digital scans.
  Unit of Measure: Millimeters (mm)

SECONDARY OUTCOMES:
Volumetric Change in Peri-Implant Tissues | Baseline (prosthesis delivery), 6 months, and annually up to 3 years post-loading
  Volumetric changes in peri-implant soft and hard tissues will be measured using 3D digital superimposition of intraoral scans. The analysis will compare changes over time in tissue volume surrounding each implant. Unit of Measure: Cubic millimeters (mm³)
Tissue Volume Difference by Crown Emergence Profile | 6 months and annually up to 3 years post-loading
  Comparison of peri-implant tissue volume changes between crowns with root-shaped apical emergence profiles versus standard crown shapes.
  Unit of Measure: Cubic millimeters (mm³)
Probing Pocket Depth at Implant Sites | 6 months and annually up to 3 years post-loading
  Probing depth at six sites per implant to evaluate peri-implant health. Unit of Measure: Millimeters (mm)
Plaque Index at Implant Sites (0-3 scale) | 6 months and annually up to 3 years
  Plaque accumulation at implant sites assessed with a modified plaque index. Unit of Measure: Score on index scale (0-3)
Bleeding on Probing at Implant Sites (percentage of sites) | 6 months and annually up to 3 years
  Presence of bleeding upon probing at six sites per implant. Unit of Measure: Percentage (%)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Sciences of Havana, Havana, Cuba

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policy and ethical considerations regarding patient confidentiality. Only aggregate-level results will be made publicly available through publications and study reports.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT07107464/Prot_SAP_000.pdf